CLINICAL TRIAL: NCT01674062
Title: An Exploratory Phase II, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Pertuzumab and Herceptin (Trastuzumab) in Patients With HER2-Positive Metastatic Breast Cancer
Brief Title: A Study of Perjeta (Pertuzumab) in Combination With Herceptin (Trastuzumab) in Participants With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO17929; 2005-003493-19 (EudraCT Number)
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Results first posted 2015-09-11 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab

ARMS (2):
- Pertuzumab + Trastuzumab (Cohorts 1 and 2) (Experimental): Females with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer will receive dual-agent treatment with pertuzumab and trastuzumab. Trastuzumab will be administered IV as 2 milligrams per kilogram (mg/kg) once weekly, or as 6 mg/kg every 3 weeks, beginning on Day 1 of Cycle 1. Pertuzumab will be administered IV at a loading dose of 840 mg followed by a standard dose of 420 mg every 3 weeks, beginning on Day 2 of Cycle 1. Thereafter, both medications will be administered on Day 1 of each 3-week cycle. Treatment will continue for a minimum of 8 cycles and may be extended until disease progression, intolerable toxicity, or death.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab
- Pertuzumab +/- Trastuzumab (Cohort 3) (Experimental): Females with HER2-positive metastatic breast cancer will receive single-agent treatment with pertuzumab. Pertuzumab will be administered IV at a loading dose of 840 mg followed by a standard dose of 420 mg every 3 weeks, administered on Day 1 of each 3-week cycle. Participants with documented disease progression may have trastuzumab added to the regimen, per the dosing schedule described for Cohorts 1 and 2, to receive dual-agent treatment until disease progression, intolerable toxicity, or death.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pertuzumab — Loading dose 840 mg IV on Day 2 of Cycle 1, followed by 420 mg every 3 weeks thereafter, until disease progression or unacceptable toxicity.
  Other Names: Perjeta
Drug: Trastuzumab — 2 mg/kg IV once weekly, or as 6 mg/kg every 3 weeks, beginning on Day 1 of Cycle 1 and on Day 1 of each 3-week cycle thereafter until disease progression or unacceptable toxicity.
  Other Names: Herceptin

SUMMARY:
This study will evaluate the efficacy and safety of Perjeta (pertuzumab) in combination with Herceptin (trastuzumab) in participants with metastatic breast cancer who have progressed on trastuzumab-based therapy (Cohorts 1 and 2), and will make a preliminary assessment of the efficacy and safety of single-agent pertuzumab (Cohort 3). Objective response rate and clinical benefit will be assessed. Pertuzumab will be administered at an initial dose of 840 milligrams (mg) intravenously (IV) on Day 1, followed by 420 mg IV every 3 weeks. Trastuzumab will be administered at the same schedule the participant was following before entry into the study. An additional cohort of participants at certain centers will receive pertuzumab monotherapy at an initial dose of 840 mg IV on Day 1, followed by 420 mg IV every 3 weeks. These participants may have trastuzumab added to the regimen in the event of progression during single-agent pertuzumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females greater than or equal to (≥) 18 years of age, with histologically-confirmed HER2-positive breast cancer
* Metastatic breast cancer, with progression on trastuzumab-based therapy as last treatment for metastatic disease
* Less than or equal to (≤) 3 chemotherapy regimens prior to study entry
* Last trastuzumab dose ≤9 weeks before study entry for participants receiving pertuzumab + trastuzumab, and ≥4 weeks for participants receiving pertuzumab monotherapy
* Left ventricular ejection fraction ≥55% at study entry

Exclusion Criteria:

* Previous treatment with an anti-cancer vaccine or any targeted therapy other than trastuzumab
* Brain metastases
* History of any cardiac adverse event related to trastuzumab therapy
* Any other malignancy in the last 5 years, except for basal cell cancer or cancer in situ of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (18):
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- France (4):
  - Besançon
  - Dijon
  - Lille
  - Montpellier
- Italy (3):
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Milan, Lombardy
- Spain (2):
  - Barcelona, Barcelona
  - Valencia, Valencia
- United Kingdom (4):
  - Edinburgh
  - Manchester
  - Northwood
  - Truro

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 99 participants with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer were screened for Cohorts 1 and 2, of whom 66 were recruited. Following primary analysis of Cohorts 1 and 2, a total of 51 new participants were screened for Cohort 3, of whom 29 were recruited.
Groups:
- Pertuzumab + Trastuzumab (Cohorts 1 and 2): Females with HER2-positive metastatic breast cancer received dual-agent treatment with pertuzumab and trastuzumab. Recruitment for Cohorts 1 and 2 was conducted separately; however, the same regimen was administered to both sets of participants. Trastuzumab was administered via intravenous (IV) infusion as 2 milligrams per kilogram (mg/kg) once weekly, or as 6 mg/kg every 3 weeks, beginning on Day 1 of Cycle 1. Pertuzumab was administered via IV infusion at a loading dose of 840 milligrams (mg) followed by a standard dose of 420 mg every 3 weeks, beginning on Day 2 of Cycle 1. Thereafter, both medications were administered on Day 1 of each 3-week cycle. Treatment continued for a minimum of 8 cycles and could be extended until disease progression, intolerable toxicity, or death.
- Pertuzumab +/- Trastuzumab (Cohort 3): Females with HER2-positive metastatic breast cancer received single-agent treatment with pertuzumab. Recruitment for Cohort 3 was conducted following primary analysis of Cohorts 1 and 2. Pertuzumab was administered via IV infusion at a loading dose of 840 mg followed by a standard dose of 420 mg every 3 weeks, administered on Day 1 of each 3-week cycle. Participants with documented disease progression could have trastuzumab added to the regimen, per the dosing schedule described for Cohorts 1 and 2, to receive dual-agent treatment until disease progression, intolerable toxicity, or death.
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2) | Pertuzumab +/- Trastuzumab (Cohort 3)
Started | 66 | 29
Completed | 0 | 0
Not Completed | 66 | 29
Not completed — Insufficient Therapeutic Response | 56 | 26
Not completed — Other | 8 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Programming Error | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Population: All randomized participants who received any amount of study medication.
Groups:
- Pertuzumab + Trastuzumab (Cohorts 1 and 2): Females with HER2-positive metastatic breast cancer received dual-agent treatment with pertuzumab and trastuzumab. Recruitment for Cohorts 1 and 2 was conducted separately; however, the same regimen was administered to both sets of participants. Trastuzumab was administered via IV infusion as 2 mg/kg once weekly, or as 6 mg/kg every 3 weeks, beginning on Day 1 of Cycle 1. Pertuzumab was administered via IV infusion at a loading dose of 840 mg followed by a standard dose of 420 mg every 3 weeks, beginning on Day 2 of Cycle 1. Thereafter, both medications were administered on Day 1 of each 3-week cycle. Treatment continued for a minimum of 8 cycles and could be extended until disease progression, intolerable toxicity, or death.
- Total: Total of all reporting groups
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2) | Pertuzumab +/- Trastuzumab (Cohort 3) | Total
Number analyzed (Participants) | 66 | 29 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.60) | 53.0 (7.95) | 54.3 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 29 | 95
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Percentage of Participants With a Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 During Dual-Agent Treatment
Description: Tumor response was assessed using RECIST version 1.0 to determine the objective response (OR) rate, or the percentage of participants with either confirmed CR or PR. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30 percent (%) decrease in the sum of the longest diameter compared to Baseline. Response was to be confirmed a minimum of 4 weeks after the initial response was documented. The OR rate was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 9.5 years (at Screening; on Day 15 of Cycles 2, 4, 6, and 8 [cycle length 3 weeks]; then every 3 months until disease progression)
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
percentage of participants | 24.2 [17.4 to 32.3]

2. Primary Outcome: Cohorts 1 and 2: Percentage of Participants With a Confirmed Best Overall Response of CR, PR, or Stable Disease (SD) According to RECIST Version 1.0 During Dual-Agent Treatment
Description: Tumor response was assessed using RECIST version 1.0 to determine the clinical benefit response (CBR) rate, or the percentage of participants with either confirmed CR or PR, or SD lasting at least 6 months. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter compared to Baseline. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient (20%) increase to qualify for disease progression, in addition to no new target lesions. Response was to be confirmed a minimum of 4 weeks after the initial response was documented. The CBR rate was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 1
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
percentage of participants | 50.0 [41.5 to 58.5]

3. Secondary Outcome: Cohort 3: Percentage of Participants With a Confirmed Best Overall Response of CR or PR According to RECIST Version 1.0 During Single-Agent Treatment With Pertuzumab
Description: Tumor response was assessed using RECIST version 1.0 to determine the OR rate, or the percentage of participants with either confirmed CR or PR. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter compared to Baseline. Response was to be confirmed a minimum of 4 weeks after the initial response was documented. The OR rate was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 7.5 years (at Screening; on Day 15 of Cycles 2, 4, 6, and 8 [cycle length 3 weeks]; then every 3 months until disease progression)
Population: All Treated Population (Cohort 3 only).
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Pertuzumab (Cohort 3): Females with HER2-positive metastatic breast cancer received single-agent treatment with pertuzumab. Recruitment for Cohort 3 was conducted following primary analysis of Cohorts 1 and 2. Pertuzumab was administered via IV infusion at a loading dose of 840 mg followed by a standard dose of 420 mg every 3 weeks, administered on Day 1 of each 3-week cycle. The treatment regimen was maintained until disease progression, intolerable toxicity, death, and/or transition to dual-agent therapy with trastuzumab.
Arm/Group | Pertuzumab (Cohort 3)
Number analyzed (Participants) | 29
percentage of participants | 3.4 [0.4 to 12.8]

4. Secondary Outcome: Cohort 3: Percentage of Participants With a Confirmed Best Overall Response of CR, PR, or SD According to RECIST Version 1.0 During Single-Agent Treatment With Pertuzumab
Description: Tumor response was assessed using RECIST version 1.0 to determine the CBR rate, or the percentage of participants with either confirmed CR or PR, or SD lasting at least 6 months. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter compared to Baseline. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient (20%) increase to qualify for disease progression, in addition to no new target lesions. Response was to be confirmed a minimum of 4 weeks after the initial response was documented. The CBR rate was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 3
Population: All Treated Population (Cohort 3 only).
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab (Cohort 3)
Number analyzed (Participants) | 29
percentage of participants | 10.3 [3.9 to 21.6]

5. Secondary Outcome: Cohorts 1 and 2: Duration of Response According to RECIST Version 1.0
Description: Tumor response was assessed using RECIST version 1.0 to determine OR and CBR rates. Duration of OR was defined as time from initial response of CR or PR to time of disease progression or death. Duration of CBR was defined similarly as time from initial response of CR or PR, or SD lasting at least 6 months, to time of disease progression or death. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter compared to Baseline. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient (20%) increase to qualify for disease progression, in addition to no new target lesions. Participants without progression or death following confirmed CR or PR were censored at the last tumor assessment. Duration of response was estimated using Kaplan-Meier analysis and expressed in weeks.
Time Frame: as for outcome 1
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
weeks
  Objective response | 40.1 [12 to 413]
  Clinical benefit response | 50.14 [12.4 to 183.7]

6. Secondary Outcome: Cohorts 1 and 2: Time to Objective Response According to RECIST Version 1.0
Description: Tumor response was assessed using RECIST version 1.0 to determine the OR rate. Time to response was defined as the time from first dose to the time of initial response of CR or PR. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter compared to Baseline. Participants with disease progression were censored at the time of progression, and those with neither disease progression nor OR were censored at the last tumor assessment. Time to response was estimated using Kaplan-Meier analysis and expressed in weeks.
Time Frame: Up to approximately 21 months (at Screening; on Day 15 of Cycles 2, 4, 6, and 8 [cycle length 3 weeks]; then every 3 months until disease progression; final analysis using February 2008 cutoff date)
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
weeks | 11.14 [4.9 to 37.3]

7. Secondary Outcome: Cohorts 1 and 2: Percentage of Participants With Disease Progression According to RECIST Version 1.0
Description: Tumor response was assessed using RECIST version 1.0 to assess for disease progression, defined as at least a 20% increase in the sum of the longest diameter, taking as reference the smallest sum of the longest diameter observed at previous tumor assessment, or the appearance of any new lesions. The percentage of participants with disease progression was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 1
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
percentage of participants | 93.9

8. Secondary Outcome: Cohorts 1 and 2: Time to Progression (TTP) According to RECIST Version 1.0
Description: Tumor response was assessed using RECIST version 1.0 to assess for disease progression, defined as at least a 20% increase in the sum of the longest diameter, taking as reference the smallest sum of the longest diameter observed at previous tumor assessment, or the appearance of any new lesions. TTP was defined as the time from first dose to the time of first documented disease progression. Participants who withdrew from the study without documented progression were censored at the last tumor assessment. TTP was estimated using Kaplan-Meier analysis and expressed in weeks.
Time Frame: as for outcome 1
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
weeks | 23.2 [4 to 244]

9. Secondary Outcome: Cohorts 1 and 2: Progression-Free Survival (PFS) According to RECIST Version 1.0
Description: Tumor response was assessed using RECIST version 1.0 to assess for disease progression, defined as at least a 20% increase in the sum of the longest diameter, taking as reference the smallest sum of the longest diameter observed at previous tumor assessment, or the appearance of any new lesions. PFS was defined as the time from first dose to the time of disease progression or death. Participants without progression or death were censored at the last tumor assessment. PFS was estimated using Kaplan-Meier analysis and expressed in weeks.
Time Frame: as for outcome 1
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Median (80% Confidence Interval); unit: weeks
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
weeks | 24.0 [18 to 34]

10. Secondary Outcome: Cohorts 1 and 2: Percentage of Participants Who Died
Description: Participants were followed for survival data during and after treatment for a maximum of 3 years after the last dose until death, withdrawal of consent, or loss to follow-up. The percentage of participants who died was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 4.5 years (during treatment; then every 4 months until death, withdrawn consent, loss to follow-up, or 3 years after last dose; final analysis using November 2010 cutoff date)
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
percentage of participants | 30.3

11. Secondary Outcome: Cohorts 1 and 2: Overall Survival (OS)
Description: Participants were followed for survival data during and after treatment for a maximum of 3 years after the last dose until death, withdrawal of consent, or loss to follow-up. OS was defined as the time from first dose to the time of death from any cause. Participants who did not experience death were censored at the last known alive date. OS was estimated using Kaplan-Meier and expressed in months.
Time Frame: as for outcome 10
Population: All Treated Population (Cohorts 1 and 2 only).
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2)
Number analyzed (Participants) | 66
months | 38.5 [32 to NA] — The value could not be calculated due to insufficient follow-up at the time the analysis was conducted.

ADVERSE EVENTS:
Time Frame: Up to approximately 9.5 years (from Day 1 until treatment discontinuation)
Description: Analysis Population Description: All Treated Population.
Arm/Group | Pertuzumab + Trastuzumab (Cohorts 1 and 2) | Pertuzumab +/- Trastuzumab (Cohort 3)
Serious Adverse Events (participants affected / at risk) | 12/66 | 1/29
Other Adverse Events (participants affected / at risk) | 62/66 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab + Trastuzumab (Cohorts 1 and 2) (N=66) | Pertuzumab +/- Trastuzumab (Cohort 3) (N=29)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Osmotic demyelination syndrome (Nervous system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Toe amputation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab + Trastuzumab (Cohorts 1 and 2) (N=66) | Pertuzumab +/- Trastuzumab (Cohort 3) (N=29)
Diarrhoea (Gastrointestinal disorders) | 42 | 16
Nausea (Gastrointestinal disorders) | 19 | 12
Vomiting (Gastrointestinal disorders) | 9 | 10
Constipation (Gastrointestinal disorders) | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 8 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4
Abdominal distension (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Stomatitis (Gastrointestinal disorders) | 6 | 0
Haemorroids (Gastrointestinal disorders) | 4 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 24 | 8
Asthenia (General disorders) | 9 | 6
Pyrexia (General disorders) | 6 | 2
Chest pain (General disorders) | 5 | 2
Chills (General disorders) | 4 | 3
Mucosal inflammation (General disorders) | 6 | 1
Influenza like illness (General disorders) | 3 | 3
Oedema peripheral (General disorders) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 18 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 8 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 5 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 15 | 4
Dizziness (Nervous system disorders) | 9 | 3
Paraesthesia (Nervous system disorders) | 8 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nasopharyngitis (Infections and infestations) | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Localised infection (Infections and infestations) | 5 | 0
Rhinitis (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 11 | 6
Insomnia (Psychiatric disorders) | 4 | 1
Weight decreased (Investigations) | 0 | 4
Left ventricular dysfunction (Cardiac disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Although the study was designed as single-arm study, as reflected in the study title, an additional cohort was opened to evaluate the efficacy and safety of single-agent pertuzumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.